CLINICAL TRIAL: NCT05834621
Title: AMNIOmics: A Prenatal Rapid Genome Validation Study
Status: Withdrawn | Type: Observational
Why Stopped: No patients were enrolled
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Myra J. Wick, Principal Investigator, Mayo Clinic
Other Study IDs: 22-002719
Record Dates: First submitted 2023-04-04; First posted 2023-04-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Multiple Anomalies of Fetus; Genetic Predisposition Suspected; Amniocentesis Affecting Fetus or Newborn; Family Members

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to validate Whole Genome Sequencing (WGS) on amniotic fluid to reduce the time to diagnosis and enhance the care for the fetus/neonate.

ELIGIBILITY:
Inclusion Criteria

* Fetus with multiple anomalies/suspected genetic disease.
* Pregnant patient already planning on having an amniocentesis for another reason separate from this study.

Exclusion Criteria

* Parents under the age of 18.
* Parents lacking the capacity to consent.
* Institutionalized (i.e., Federal Medical Prison).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be identified internally through provider referrals most commonly through the Mayo Clinic Obstetrical and Maternal Fetal Medicine services.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Validation of Rapid Whole Genome Sequencing technology on amniotic fluid samples | 5 years
  Collection of both amniotic fluid and blood samples to compare results of whole genome sequencing for a fetus with suspected genetic disease.
Enrollment of study participants | 5 years
  To recruit up to 90 total participants including child and both parents
Collection of Biospecimens | 5 years
  Total number of biospecimens collected which may include both blood samples and amniotic fluid

CONTACTS AND LOCATIONS:
Overall Officials: Myra Wick, MD, PhD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials